CLINICAL TRIAL: NCT01994369
Title: A Pilot & Feasibility Study of the Imaging Potential of EC17 in Subjects Undergoing Surgery Presenting Breast Cancer
Brief Title: Intraoperative Imagery of Breast Cancer With Folate-FITC (EC17)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sunil Singhall, Assistant Professor of Medicine, Assistant Professor of Surgery, Director Thoracic Surgery Research Laboratory, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 818065; 818065 [UPenn IRB Protocol#]
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Resectable Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EC17 Injection group (Experimental): This group with receive a single dose of EC17, infused over 10 minutes, prior to surgery. Then, during surgery, they will be imaged with a camera and an imaging probe the investigators have developed.
  Interventions: Drug: EC17

INTERVENTIONS:
Drug: EC17
  Other Names: Folate-FITC

SUMMARY:
Breast cancer is the most common cancer and the second cause of cancer mortality in women. There are approximately 200,000 new cases of breast cancer a year. Classically, breast cancers are divided into two groups, invasive and non-invasive. A mainstay of the treatment of both of these types is surgical resection not only for therapeutic purposes but also for diagnostic purposes. Breast conserving therapy includes surgical lumpectomy and post-operative radiation. However, despite best surgical practices, when patients undergo BCT anywhere from 20 - 40% of these patients have margins positive for cancer. This leads to increased rates of reoperation which are quoted to be as high as 30% and increased local recurrences.

There is an over expression of folate receptors located on the surface of many human carcinoma nodules.Specifically for breast cancer up to 33% of all breast cancers over express the folate receptor.

Folate-fluorescein isothiocyanate, or folate-FITC, also identified as EC-17, targets folate receptors over expressed in certain cancers such as breast cancer, and could help in better identifying the margins of the cancer thereby achieving negative margins.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years of age and older
2. Patients presenting with breast cancer presumed to be resectable by lumpectomy and/or mastectomy on pre-operative assessment
3. Good operative candidate
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

1. Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery
2. Patients with a history of anaphylactic reactions to Folate-FITC or insects
3. At-risk patient populations

   1. "People who would be easily lost to follow up (ex: People who are homeless or alcohol dependent)
   2. Patients unable to participate in the consent process (children and neonates).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The ability of EC17 and the imaging system to detect FRA positive tumors during surgery conducted 2-4 hours post EC-17 administration. | Within two to four hours of injection of EC17

SECONDARY OUTCOMES:
The number of participants that will have an adverse reaction to the EC17 | Day 1- Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States